CLINICAL TRIAL: NCT03287557
Title: Dysregulated CNS Inflammation After Acute Brain Injury
Status: Completed | Type: Observational
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Linda Van Eldik, Sponsor Investigator, University of Kentucky
Other Study IDs: 17-0583-F6A
Record Dates: First submitted 2017-09-12; First posted 2017-09-19 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Traumatic Brain Injury; Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CSF will be collected from an external ventricular drain (EVD) at five time points post-injury: 6, 12, 24, 48, 60 hrs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
By doing this study, the investigator hopes to learn how the levels of important proteins involved in inflammation change over time in patients with acute brain injury. The total amount of time participants will be asked to volunteer for this study is approximately two hours over a five day period.

DETAILED DESCRIPTION:
This pilot project is a prospective, observational study in 20 patients who are admitted to University of Kentucky (UK) Chandler Medical Center with a diagnosis of severe, non-penetrating traumatic brain injury (TBI) or aneurysmal subarachnoid hemorrhage (aSAH).

All adult participants with a primary diagnosis of severe, non-penetrating TBI or aSAH who are admitted to the neuroscience or trauma intensive care units will be screened for potential inclusion into this study. Once a potential participant is identified, the legally-authorized representative will be approached for study consent and HIPAA authorization. If the participant regains consent capacity before the end of the cerebrospinal fluid (CSF) collection period, assent will be obtained from the research participant.

In this research study, up to 5 small samples of CSF, will be carefully removed from the device, already in place, that drains excess CSF from the participant's head. The samples will be less than 1 teaspoon (< 5 mL) each. These samples will be frozen and stored until samples from approximately 20 participants have been obtained.

These samples will then be prepared and sent to a research laboratory to analyze the proteins in the samples collected from each research participant.

Because the results of this study will not affect the treatment participants receive in or outside of the hospital, the investigator will not share the results of this study with the participant, their doctor or their family member(s).

ELIGIBILITY:
Inclusion Criteria:

* severe, non-penetrating TBI or aSAH
* must have a ventriculostomy (EVD) placed by the UK Neurosurgery service within 12 hours of primary traumatic episode

Exclusion Criteria:

* non-survivable brain injury or other organ system injury
* life expectancy is five days or less
* penetrating TBI
* status epilepticus upon arrival to the hospital
* severe ischemic heart disease or congestive heart failure, myocardial infarction, or spinal cord injury
* Takotsubo cardiomyopathy secondary to the SAH
* active cancer or have been treated for cancer within the previous 6 months

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants selected will come from those who have been admitted to the University of Kentucky (UK) medical center
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Severe TBI - Measure of temporal profile of inflammatory proteins in CSF | For 24 months from start of the study
  CSF collection

SECONDARY OUTCOMES:
aSAH - Measure of temporal profile of inflammatory proteins in CSF | For 24 months from start of the study
  CSF collection

CONTACTS AND LOCATIONS:
Overall Officials: Linda J Van Eldik, PhD, Study Director — University of Kentucky
Locations (1):
- University of Kentucky Deparment of Neurosurgery, UK Chandler Hospital, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No